CLINICAL TRIAL: NCT01200342
Title: Phase II Study of Genasense-Carboplatin-Paclitaxel-Combination in Uveal Melanoma
Brief Title: Genasense, Carboplatin, Paclitaxel (GCP) Combination in Uveal Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical company no longer manufacturing investigational product.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0188
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Melanoma
Keywords: Uveal melanoma; Carboplatin; Genasense; Paclitaxel; oblimersen; GCP
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — oblimersen; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genasense + Paclitaxel + Carboplatin (Experimental): Genasense 900 mg intravenous (IV) on a fixed-dose as a 1-hour infusion on Days 1, 3, and 5 of a 21 day cycle; Paclitaxel 175 mg/m^2 IV over 3 hours Day 3 after Genasense; Carboplatin dose in mg (target area under the concentration [AUC)]=6) administered over 30 minutes IV Piggyback (IVPB) on Day 3 after Paclitaxel.
  Interventions: Drug: Genasense; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Genasense — 900 mg by vein over 1 hour on Days 1, 3, and 5 of a 21 day cycle.
  Other Names: G3139; Oblimersen
Drug: Paclitaxel — 175 mg/m^2 by vein over 3 hours on Day 3 of a 21 day cycle following Genasense.
  Other Names: Taxol
Drug: Carboplatin — Carboplatin starting dose in mg (AUC= 6) is administered over 30 minutes IV Piggyback (IVPB). Carboplatin will be dosed after Paclitaxel dose on Day 3 every 3 weeks.
  The total dose of Carboplatin is calculated using a formula based upon a participant's glomerular filtration rate (GFR in mL/min) and Carboplatin target area under the concentration (AUC).
  Other Names: Paraplatin

SUMMARY:
The goal of this clinical research is to learn if the combination of Genasense (oblimersen), carboplatin, and paclitaxel (GCP) can help to control metastatic uveal melanoma. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

Oblimersen is designed to stop the body from making a protein that makes melanoma cells resistant to chemotherapy drugs. This may make carboplatin and/or paclitaxel more effective.

Carboplatin is designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

Paclitaxel is designed to block cancer cells from dividing, which may cause them to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive oblimersen by vein over about 1 hour (+/- 5 minutes) on Days 1, 3, and 5 of each 21-day study "cycle." You will receive dexamethasone by vein over about 30 minutes before you receive oblimersen to help prevent side effects. You will take ibuprofen by mouth about 30 minutes before you receive oblimersen.

You will receive paclitaxel by vein over about 3 hours (+/- 5 minutes) on Day 3 of each cycle.

You will receive carboplatin by vein over about 30 minutes (+/- 5 minutes) on Day 3 of each cycle.

Before you receive each of these drugs, you may receive other drugs to help prevent side effects (such as nausea, vomiting, fever, and/or body aches). You may need to receive some of these drugs for some time after you receive the study drugs. Your doctor will tell you more about each of these drugs, about how they are given, and about any possible risks of receiving them.

Study Visits:

Within 3 days before each cycle, blood (about 1 tablespoon) will be drawn for routine tests.

On Day 1 of each cycle:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any side effects you may be having.
* Women who are able to become pregnant will have a routine urine pregnancy test done.

Each week while you are on study, blood (about 1 teaspoon) will be drawn for routine tests.

Every 6 weeks, you will have the same imaging (CT and/or MRI) scans that you had at screening to check the status of the disease. If the doctor thinks it is needed, you will have a bone scan.

Length of Study:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over once you have completed the end-of-treatment visit and follow-up.

End-of-Treatment Visit:

After you stop receiving the study drugs, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will be asked about any side effects you may have had.
* You will have the same imaging (CTand /or MRI) scans that you had at screening to check the status of the disease.
* Women who are able to become pregnant will have a routine urine pregnancy test done.

Follow-up:

Every 3 months for up to 2 years after you stop receiving the study drugs, you will be called and asked about how you are doing and about any other drugs you may be receiving. Each call will last about 3 minutes.

This is an investigational study. Carboplatin and paclitaxel are FDA approved and commercially available for the treatment of a variety of cancers including breast, lung, and ovarian cancers. Oblimersen is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a history of uveal melanoma and documented metastatic disease
2. Patients must have at least one measurable lesion as per revised RECIST Criteria. A measurable lesion is defined as a non-nodal lesions that is >/= 10 mm provided the CT slice is </=5 mm in thickness or a pathologic lymph node that is >/= 15 mm on the short axis provided the CT slice is </= 5 mm in thickness or Superficial skin lesion that is >/= 10 mm in diameter as assessed using calipers. Bone lesions are not considered measurable.
3. Patients may be previously untreated or may have received prior systemic therapy but no more than one systemic cytotoxic chemotherapy regimen and one targeted therapy for metastatic disease.
4. At least 6 weeks (42 days) since any prior immunotherapy, cytokine, biologic, vaccine or other therapy unless patients have progressed during therapy. If progression occurred during therapy, patient must have recovered from any side effects before starting GCP therapy.
5. At least 4 weeks (28 days) since prior radiotherapy to > 20% of the bone marrow.
6. Lesions being used to assess disease status may not have been radiated or if so, must have progressed during or after radiation therapy.
7. Patients must have ECOG performance status of 0 - 2.
8. Patients should be 18 years of age or older.
9. Patients must have adequate liver and renal function as defined by total bilirubin </=1.5 mg/dl, serum Lactate Dehydrogenase level no higher than 2.0 x UNL of the institution, transaminase (i.e., ALT and AST) levels no higher than 5 x UNL and serum creatinine </=1.5 mg/dl or estimated Creatinine Clearance >/=60 ml/min
10. Patients must have adequate bone marrow function as defined by an absolute neutrophil count of greater or equal to 1,500/mm3, and platelet count of greater or equal to 100,000/mm3.
11. Patients must sign an informed consent form indicating that they are aware of the investigational nature of this study and in keeping with the policies of the institution.
12. Females of childbearing potential (non childbearing is defined as greater than one year post-menopausal or surgically sterilized) must use acceptable contraceptive methods (abstinence, intrauterine device, oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 7 days prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study.

Exclusion Criteria:

1. Patients who have received prior therapy with Genasense, any taxane or any of cisplatin analogues for systemic disease.
2. Patients whose site of primary melanoma is not in the choroid.
3. Patients who have a current history of neoplasm other than the entry diagnosis, except for curatively treated non-melanoma skin cancer or carcinoma in situ of the prostate or cervix or other cancers treated for cure and with a disease-free survival longer than 2 years.
4. Patients with brain metastasis or history of brain metastasis (es).
5. Patients who are pregnant or breastfeeding.
6. Patients with current active infections requiring anti-infectious treatment (e.g., antibiotics, antivirals, or antifungals).
7. Patients with current peripheral neuropathy of any etiology that is greater than grade one (1).
8. Patients with unstable or serious concurrent medical conditions are excluded. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent. PI or his designee shall make the final determination regarding appropriateness of enrollment.
9. Patients with a known hypersensitivity to cremophor containing anti-cancer agents.
10. Patients with one or more of the following as the only manifestations of disease are ineligible: Osteoblastic bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, carcinomatous lymphangitis, CNS metastases, lesions in a previously irradiated area that have not shown definite progression, or disease only inferred from laboratory tests or markers.
11. Patients with Gilbert's Syndrome.
12. Patients must not have had major surgery within the past 14 days.
13. Patients must not receive any concurrent chemotherapy, radiotherapy, or immunotherapy while on study.
14. Known HIV disease or infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sapna P. Patel, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 6, 2010 to November 05, 2012. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Study was terminated early due to decision by drug sponsor to no longer manufacture investigational drug.
Period: Overall Study
Arm/Group | Genasense + Paclitaxel + Carboplatin
Started | 7
Completed | 6
Not Completed | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Population: Due to inadequate enrollment of study participants, no statistical analysis were able to be performed.
Arm/Group | Genasense + Paclitaxel + Carboplatin
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 61 [61 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Percentage Subjects With Confirmed Complete or Partial Response)
Description: Tumor response by Response Evaluation Criteria in Solid Tumors for participants with measurable disease defined by presence of at least 1 measurable lesion at baseline: Complete Response (CR): disappearance all target lesions determined by 2 consecutive observations not less than 4 weeks apart. Partial Response (PR): >30% decrease in sum of LD of target lesions (LD) of target lesions taking as reference baseline sum LD determined by two consecutive observations not less than four weeks apart. Progression (PD): >20% increase in sum of LD of target lesions references smallest sum LD recorded since treatment started or appearance of one or more new lesions. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking references smallest sum LD since treatment started. Measurable: lesions accurately measured in at least 1 dimension (longest diameter to be recorded) as 20 mm with conventional techniques or as 10 mm with spiral CT s
Time Frame: Following two 3-week cycles
Population: The efficacy-evaluable population defined as all subjects who completed at least two cycles of therapy and had at least one post-screening assessment of target and non-target lesions. Due to inadequate enrollment of study participants, no statistical analyses were able to be performed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Genasense + Paclitaxel + Carboplatin
Number analyzed (Participants) | 7
Percentage of Participants | 0

2. Primary Outcome: Number of Participants With Response
Description: as for outcome 1
Time Frame: Following two 3-week cycles
Population: The efficacy-evaluable population defined as all subjects who completed at least two cycles of therapy and had at least one post-screening assessment of target and non-target lesions.
Measure: Number; unit: Participants
Arm/Group | Genasense + Paclitaxel + Carboplatin
Number analyzed (Participants) | 7
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Progressive Disease (PD) | 1
  Stable Disease (SD) | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the day of initial treatment with study drug until thirty (30) days after the last treatment.
Description: Collection Period: April 01, 2011 to September 06, 2013.
Arm/Group | Genasense + Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genasense + Paclitaxel + Carboplatin (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 2 (2)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 4 (4)
Alopecia (General disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 5 (10)
Anorexia (Psychiatric disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 3 (3)
Blood bilirubin increased (Blood and lymphatic system disorders) | 2 (2)
Blurred vision (Eye disorders) | 2 (2)
Chills (General disorders) | 4 (4)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6) — 1 event = Grade 3
Cough (General disorders) | 2 (3)
Creatinine increased (Renal and urinary disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (10)
Dizziness (Ear and labyrinth disorders) | 4 (6) — 1 event = Grade 3
Dry mouth (General disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Edema limbs (Musculoskeletal and connective tissue disorders) | 1 (2)
Eye disorders (Eye disorders) | 1 (3)
Fatigue (General disorders) | 6 (12) — 1 event = Grade 3
Febrile neutropenia (Infections and infestations) | 1 (1) — Grade 3
Fever (Infections and infestations) | 2 (2)
Gait disturbance (Nervous system disorders) | 1 (1) — Loss of balance
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Hallucinations (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hot flashes (General disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 4 (6) — 2 events = Grade 3; 1 event = Grade 4
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Hyperuricemia (Renal and urinary disorders) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (2)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 3 (6) — 1 event = Grade 3
Hypotension (Cardiac disorders) | 1 (1) — Grade 3
Infections and infestations (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Immune system disorders) | 5 (8)
Mucositis oral (Infections and infestations) | 2 (5)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (General disorders) | 6 (13)
Neutrophil count decreased (Immune system disorders) | 4 (12) — 2 events = Grade 3; 2 events = Grade 4
Pain (General disorders) | 1 (1) — l.thorax
Pain (General disorders) | 1 (1) — lower back
Pain (General disorders) | 1 (1) — Abdominal
Pain (General disorders) | 1 (1) — gr. 1 BL pain
Pain (General disorders) | 1 (2) — joint pains
Pain (General disorders) | 2 (4) — 1 event = Grade 3
Pain (General disorders) | 1 (1) — sharp joint pains
Pain (General disorders) | 1 (1) — Lt nares through eye
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Musculoskeletal and connective tissue disorders) | 7 (9)
Platelet count decreased (Blood and lymphatic system disorders) | 6 (12) — 1 event = Grade 3
Pruritus (Infections and infestations) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 (3)
Skin infection (Infections and infestations) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2) — 1 event = Grade 3
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Vascular disorders (Vascular disorders) | 1 (1)
Vomiting (General disorders) | 6 (10) — 1 event = Grade 3
Weight loss (General disorders) | 2 (3)
White blood cell decreased (Immune system disorders) | 4 (8) — 3 events = Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes